CLINICAL TRIAL: NCT02867319
Title: Safety Study of ACYW135 Meningococcal Polysaccharide Vaccine Aged 2-50 Years Old
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Chaoyang District Centre for Disease Control and Prevention (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: cycdc2016-3
Record Dates: First submitted 2016-08-11; First posted 2016-08-15 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Meningococcal
Keywords: safety; vaccine

ARMS (3):
- age of 18-50 years old (Experimental)
  Interventions: Biological: A dose of ACYW135 meningococcal polysaccharide vaccine
- age of 7-17 years old (Experimental)
  Interventions: Biological: A dose of ACYW135 meningococcal polysaccharide vaccine
- age of 2-6 years old (Experimental)
  Interventions: Biological: A dose of ACYW135 meningococcal polysaccharide vaccine

INTERVENTIONS:
Biological: A dose of ACYW135 meningococcal polysaccharide vaccine — A dose of ACYW135 meningococcal polysaccharide vaccine will be given in certain arm.

SUMMARY:
This phase I clinical study evaluates the safety of ACYW135 meningococcal polysaccharide vaccine in population aged 2-6, 7-17, 18-50 years old by the method of both passive and active surveillance.

ELIGIBILITY:
Inclusion Criteria:

* With the subject (or his guardian's) informed consent and signed the informed consent;
* The history, physical examination and clinical judgement were determined to be healthy and in accordance with the vaccination age of the product;
* The Subject or his guardian could comply with the clinical study protocol;
* Have not been inoculated with Meningococcal vaccine in the past six months and A + C meningococcal polysaccharide vaccine in the past two years;
* Have not been inoculated with other preventive biological products;
* Axillary temperature≤37.0 ℃.

Exclusion Criteria:

* Children with the history of Neisseria meningitis;
* Had allergies or serious adverse reactions of previous vaccination, such as allergies, urticaria, dyspnea, edema, abdominal pain, etc;
* Had immune inhibitor therapy and cytotoxic therapy, inhaled corticosteroids in the past 6 months (not including allergic rhinitis corticosteroid aerosol therapy, patients with acute non concurrent dermatitis surface corticosteroid therapy);
* Have been accepted blood products in the past 3 months;
* Have been inoculated with other research drugs or vaccines in the past month;
* Have been inoculated with attenuated live vaccine in the past 14 days;
* Have been inoculated with subunit or inactivated vaccine in the past 7 days;
* Had any acute illness, the need for systemic application of antibiotics or antiviral treatment in the past 7 days;
* Had fever in the past 3 days (axillary temperature≥38.0℃) ;
* Have been diagnosed with abnormal coagulation function (such as the lack of coagulation factors, coagulation disorders and abnormal blood platelet), obvious bruises or coagulation disorders by physician diagnosis;
* Had the history of thyroid resection or the need for treatment of thyroid diseases in the past 12 months;
* Asplenia, functional asplenia and asplenia or splenectomy of any situation;
* Had epilepsy, convulsions, encephalopathy, mental illness or family history;
* Suffering from serious chronic diseases (such as Down's syndrome, diabetes, sickle cell anemia, neurological disorders or Guillain-Barre syndrome);
* Suffering from known or suspected concurrent diseases including: respiratory diseases, acute or chronic infection of the activities, children's mother or the subject had HIV infection, cardiovascular disease, high blood pressure, during cancer treatment period, skin diseases;
* The female during her pregnant and lactation period or who plan to become pregnant during the trial.
* The subject of any other factors that are not suitable to participate in clinical trials according to the researcher's judgment.

Ages: 2 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2016-03; Primary Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
The rate of adverse reactions of ACYW135 meningococcal polysaccharide vaccine | 28 days
  Adverse reactions associated with vaccine will be observed in subjects after each vaccination. Solicited local adverse events include Pain, Redness, Swelling, Induration, Rash, Pruritus at injection site. solicited general adverse events include Fever, Nausea, Vomiting, Diarrhea, Decreased appetite, Be agitated (irritability, abnormal crying), fatigue, allergy